CLINICAL TRIAL: NCT04710394
Title: Efficacy of Bimodal Visual-Olfactory Training in Participants With COVID-19 Resultant Hyposmia or Anosmia Using Participant-Preferred Scents
Brief Title: Visual-OLfactory Training in Participants With COVID-19 Resultant Loss of Smell
Acronym: VOLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 7011897206
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Anosmia; Covid19; Ageusia; Hyposmia; Hypogeusia; SARS-CoV-2 Infection; COVID-19 Pandemic
Keywords: Anosmia; Loss of Smell; Loss of Taste; Hyposmia; Ageusia; Covid-19; SARS-CoV-2
MeSH Terms: conditions — Anosmia; COVID-19; Ageusia | interventions — Olfactory Training

STUDY DESIGN:
Intervention Model Description: Two-by-two factorial interventional study design will lend to achieving the study aims. Participants meeting eligibility criterion will be randomized to one of four arms:
  1. Unimodal Olfactory Training with Conventional Odors
  2. Unimodal Olfactory Training with Patient-Preferred Odors
  3. Bimodal Visual, Olfactory Training with Conventional Odors
  4. Bimodal Visual, Olfactory Training with Patient-Preferred Odors
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Unimodal Olfactory Training with Conventional Odors (Active Comparator): Participants will undergo smell training without a visual component, and train using 4 pre-determined scents: rose, lemon, eucalyptus, and clove.
  Interventions: Behavioral: Smell Training
- Unimodal Olfactory Training with Patient-Preferred Odors (Experimental): Participants will undergo smell training without a visual component, and undergo an odor selection process in which they choose four scents to train with that they identify as important. A total of 24 scents will be included for patients to select from, including: Lemon, Orange, Grapefruit, Lime, Eucalyptus, Peppermint, Spearmint, Tea Tree, Rose, Lavender, Jasmine, Geranium, Frankincense, Cedarwood, Juniper, Sandalwood, Black Pepper, Oregano, Rosemary, Clove, Vanilla, Coffee, Cinnamon, Nutmeg.
  Interventions: Behavioral: Smell Training
- Bimodal Visual, Olfactory Training with Conventional Odors (Experimental): Participants will undergo smell training while simultaneously focusing on a picture of the odor, and train using 4 pre-determined scents: rose, lemon, eucalyptus, and clove.
  Interventions: Behavioral: Smell Training
- Bimodal Visual, Olfactory Training with Patient-Preferred Odors (Experimental): Participants will undergo smell training while simultaneously focusing on a picture of the odor, and undergo an odor selection process in which they choose four scents to train with that they identify as important. A total of 24 scents will be included for patients to select from, including: Lemon, Orange, Grapefruit, Lime, Eucalyptus, Peppermint, Spearmint, Tea Tree, Rose, Lavender, Jasmine, Geranium, Frankincense, Cedarwood, Juniper, Sandalwood, Black Pepper, Oregano, Rosemary, Clove, Vanilla, Coffee, Cinnamon, Nutmeg.
  Interventions: Behavioral: Smell Training

INTERVENTIONS:
Behavioral: Smell Training — Participants will be provided with 4 labeled jars, each containing an odor pre-impregnated cotton pad. Participants will sniff each scent for 10 seconds, twice daily, once in the morning and once in evening. The participant will take 30 seconds of rest between each scent. All participants will undergo this smell training regimen for 12 weeks.
  Other Names: Olfactory Training

SUMMARY:
Olfactory dysfunction is a defining symptom of COVID-19 infection. As the number of total, confirmed COVID-19 cases approached 19 million in the United States, it is estimated that there will be 250,000 to 500,000 new cases of chronically diminished smell (hyposmia) and loss of smell (anosmia) this year. Olfactory dysfunction is proposed to worsen numerous common co-morbidities in patients and has been shown to lead to a decreased quality of life. There are very few effective treatments for hyposmia or anosmia, and there is no gold standard of treatment.

One proposed treatment option is smell training, which has shown promising yet variable results in a multitude of studies. It garners its theoretical basis from the high degree of neuroplasticity within the olfactory system, both peripherally and centrally. However, due to a relative inadequacy of proper studies on olfactory training, it is unknown what the most efficacious method in which to undergo the training is. This study proposes two novel procedural modifications to smell training in an attempt to enhance its efficacy. The investigators propose using a bimodal visual-olfactory approach, rather than relying on olfaction alone, during smell training, as well as using patient-preferred scents in the training that are identified as important by the study participant, rather than pre-determined scents with inadequate scientific backing. The investigators hypothesize that by utilizing bimodal visual-olfactory training and patient-selected scents, the olfactory training will be more efficacious and more motivating for participants.

DETAILED DESCRIPTION:
Over 200,000 people visit physicians yearly for taste and smell disorders and given the well-documented prevalence of olfactory dysfunction in COVID-19 infection, there is likely to be an increased need to address these concerns. The loss of the sense of smell has been shown to be linked to decreased quality of life, depression, decreased enjoyment of the flavor of foods, and may even be a contributing factor in the physiologic anorexia of aging.

Some of the most common causes of olfactory dysfunction include post-infectious, post-traumatic, and neurodegenerative. Of these, post-viral olfactory dysfunction is the leading cause, accounting for an estimated 18.6 to 42.5% of individuals with olfactory dysfunction. Respiratory viruses found to be responsible for olfactory loss include common respiratory viruses including rhinovirus, coronavirus, parainfluenza virus, adenovirus, and influenza virus. It is then no surprise, that olfactory dysfunction is a defining symptom of COVID-19 infection. Estimates for the prevalence of smell dysfunction in COVID-19 infection vary. In a cross-sectional survey of 59 patients with COVID-19, 34% (20/59) self-reported a smell and/or taste disorder. In a multi-center European study, 85.6% (357/417) of cases with confirmed COVID-19 experienced olfactory dysfunction. Only an estimated 44% of these patients experienced recovery of olfaction after 2 weeks of convalescence from COVID-19 infection. Although it is impossible to know the long-term recovery rates of this newly emerging pathogen, as the total number of confirmed COVID-19 cases approaches 19 million in the United States, unpublished data generated by Amish Mustafa Khan in Dr. Jay F. Piccirillo's lab at Washington University estimates nearly 250,000 to 500,000 new cases of chronic olfactory dysfunction.

There is no gold standard set of guidelines for the diagnosis and treatment of post-viral hyposmia or anosmia. Most evidence for pharmacological interventions is weak, with very few controlled studies that account for spontaneous improvement overtime. Moreover, treatments that are effective for sino-nasal disease such as topical corticosteroids are not effective for sensorineural post-viral olfactory loss. A systemic review of post-viral olfactory dysfunction studied eight commonly utilized pharmacological treatments: Oral corticosteroids, local corticosteroids, zinc sulfate, alpha-lipoic acid, caroverine, Vitamin A, Gingko Bilboa, Minocycle. Improvement was noted for study participants receiving oral corticosteroids, local corticosteroids, alpha lipoid acid, and caroverine. However, these studies were of poor quality, and the authors conclude that there is no strong evidence supporting the use of any pharmacological intervention for the treatment of post-viral olfactory dysfunction.

One proposed treatment shown to be beneficial for a wide variety of etiologies of olfactory dysfunction, including post-viral upper respiratory infection, is olfactory training. The theoretical basis for olfactory training emerges from multiple experimental and clinical studies suggesting that the olfactory pathway has neuroplasticity to recover, both peripherally, due to the regenerative capacity of olfactory receptor cells, and centrally. In a study using fMRI after olfactory training, there were increased functional connections in olfactory areas such as the anterior entorhinal cortex, inferior prefrontal gyrus, and the primary somatosensory cortex, suggesting that the olfactory pathways are capable of reorganization with training. In another study, increased exposure by anosmic participants to androstenone resulted in an increase in amplitude of the olfactory evoked potential and the olfactory event-related potential, suggesting that that the peripheral olfactory receptor cells are also neuroplastic, likely due to an increase in expression of olfactory neuron receptors in response to training.

The investigators believe that patients experiencing olfactory dysfunction secondary to COVID-19 are especially good candidates for olfactory training for two reasons. Firstly, the pathophysiology of COVID-19 olfactory dysfunction is mediated through damage to the peripheral olfactory receptor cells located in the nasal epithelium lining the nasal cavity and central pathways via neuro-invasion through the olfactory pathway. This suggests that interventions most likely to be efficacious in this patient population target both central and peripheral pathways, as olfactory training does. Secondly, relative to other causes of olfactory dysfunction, post-viral olfactory dysfunction more commonly presents with hyposmia, rather than anosmia. Residual olfactory function is an important prognosticator that improves the likelihood of improvement. Furthermore, patients with post-viral olfactory dysfunction more commonly present with concurrent dysosmia than other common causes of olfactory dysfunction. It is likely that dysomia may be a result of disordered axonal regeneration. This further suggests that patients with post-viral olfactory loss are most likely to benefit from olfactory training.

Olfactory training typically consists of a patient smelling a scented oil dropped in a labeled jar on a cotton ball for a specified length of time a certain number of times per day. The details of the most efficacious method for olfactory training is not yet described, with various studies adjusting the length of time of training, frequency of training, or even adding nasal corticosteroids alongside olfactory training. While olfactory training is promising, these inconsistencies highlight the inadequacies in the training. Two unstudied areas include the effects of a bimodal visual-olfactory approach to olfactory training as well as the effects of patient preference in determining the scents in which to undergo the training.

Bimodal training has been shown to be effective in other sensory training, such as through audio-visual training to enhance the auditory adaptation process, and even in animal studies with ferrets with bilateral cochlear implants, improving auditory spatial processing. Loss of hearing has been shown to result in improved vision, adding to the hypothesis that an intimate connection exists between senses and that its relationship is worthy of continued modulation and study. Furthermore, perhaps many patients have undergone olfactory training with scents that patients have no interest in being able to smell, and perhaps patient compliance has been an underreported cause of the variability in olfactory training results due to the resulting decreased motivation to smell scents patients have no desire to be able to smell. The original clinical trial on olfactory training, and most since, have chosen to evaluate the efficacy of olfactory training using four pre-determined scents: rose (flowery), lemon (fruity), eucalyptus (resinous), and cloves (aromatic). These scents were chosen due to the work of German psychologist Hans Henning who categorized smells into six different categories: floral, putrid, fruity, burned, spicy, and resinous. The unpleasant smells of putrid and burned were omitted from the olfactory training protocol, resulting in the four smells that are often studied today. Although humans respond to odors as members of odor categories, there is little scientific basis behind making these four specific scents the standard for olfactory training. There are various studies that have used select scents or an array of other scents, however, there are no known studies that have used patient preference in choosing scents in which to undergo olfactory training.

The investigators hypothesize that using patient preference in choosing the scents that the participant is to undergo olfactory training and adding in a visual component to the training will not only be a patient-centered research approach, but also a more effective means of improving olfactory function.

ELIGIBILITY:
Inclusion Criteria:

- Subjective or clinically diagnosed olfactory dysfunction of 3 months duration or longer initially diagnosed within 2 weeks of a COVID-19 infection

Exclusion Criteria:

* Diagnosed olfactory dysfunction due to head trauma
* Chronic rhinosinusitis
* Congenital olfactory dysfunction
* Nasal polyps
* Neurodegenerative disorders (for example, Alzheimer or Parkinson Disease)
* Pre-Assessment UPSIT score ≥34 for males and ≥35 for females
* Pregnant
* Inability to read, write, and understand English
* Inability to perform home olfactory training (for example, due to limited access to internet)
* Residence outside of the the United States of America
* Previously conducting smell training

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
University of Pennsylvania Smell Identification Test (UPSIT) | Measurement will be taken at time zero (pre-intervention) and 12 weeks (post-intervention)
  The UPSIT includes 4 odor-impregnated booklets that contain 10 forced-choice multiple choice questions each for participants to scratch-and-sniff to identify various odors and is a commercially available test. Normosmia is defined as ≥34 for males and ≥35 for females, and a change of 4 points or more from baseline indicates a clinically meaningful result.

SECONDARY OUTCOMES:
Clinical Global Impression Severity (CGI-S) Scale | Measurement will be taken at time zero (pre-intervention) and 12 weeks (post-intervention)
  The CGI-S is a subjective rating scale in which a participant can rate the severity of their dysfunction. The scale is rated from 1-7 with 1 being normal sense of smell, 4 being moderate loss of smell, and 7 being complete loss of smell. Each rating has a definition to better elucidate what any particular rating might mean, so as to decrease variability between patient responses with the same subjective level of dysfunction or improvement.
Clinical Global Impression Improvement (CGI-I) Scale | Measurement will be taken at time zero (pre-intervention) and 12 weeks (post-intervention)
  The CGI-I is a subjective rating scale in which a participant can rate the rate the improvement (or lack thereof) of their dysfunction after smell training. The scale is rated from 1-7 with 1 being very much improved sense of smell, 4 being no change in sense of smell, and 7 being very much worse sense of smell. Each rating has a definition to better elucidate what any particular rating might mean, so as to decrease variability between patient responses with the same subjective level of dysfunction or improvement.
Olfactory Dysfunction Outcomes Rating (ODOR) | Measurement will be taken at time zero (pre-intervention) and 12 weeks (post-intervention)
  A 28-item health-related quality of life instrument specific for olfactory dysfunction developed by Dr. Jake Lee in Dr. Jay F. Piccirillo's lab at Washington University.

CONTACTS AND LOCATIONS:
Overall Officials: Jay F. Piccirillo, M.D., FACS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine in Saint Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and research resources generated from this clinical trial will be made available by request, while safeguarding the privacy of participants in accordance with NIH policy and HIPAA guidelines.
  The data to be shared will include information about the project, protocol, data dictionary, and the final individual de-identified research subject data. These data will include the responses to the baseline and post-intervention Olfactory Dysfunction Outcomes Rating (ODOR), Clinical Global Impression Severity (CGI-S) Scale , University of Pennsylvania Smell Identification Test (UPSIT), post-intervention Clinical Global Impression Improvement (CGI-I) Scale, and treatment assignment.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be made available within 12 months of the completion date of the research project, for 2 subsequent years.
Access Criteria: Data access will be arranged through a data-sharing agreement, which will indicate the criteria for data access, documentation of IRB approval from requestor's institution, incorporation of appropriate privacy and confidentiality standards to ensure data security at the recipient site, and prohibit manipulation of data for the purposes of identifying subjects or redistribution to third parties. Data access will be managed by the Research Compliance and Recruitment Coordinator, and data maintenance will be managed by the Study Biostatistician.
URL: http://otolaryngologyoutcomesresearch.wustl.edu/

REFERENCES:
- [Background] Runnebaum B, Runnebaum H, Stober I, Zander J. Progesterone 20 alpha-dihydroprogesterone and 20 beta-dihydroprogesterone levels in different compartments from the human foeto-placental unit. Acta Endocrinol (Copenh). 1975 Nov;80(3):558-68. doi: 10.1530/acta.0.0800558. PMID 1242570
- [Background] Croy I, Nordin S, Hummel T. Olfactory disorders and quality of life--an updated review. Chem Senses. 2014 Mar;39(3):185-94. doi: 10.1093/chemse/bjt072. Epub 2014 Jan 15. PMID 24429163
- [Background] Neuland C, Bitter T, Marschner H, Gudziol H, Guntinas-Lichius O. Health-related and specific olfaction-related quality of life in patients with chronic functional anosmia or severe hyposmia. Laryngoscope. 2011 Apr;121(4):867-72. doi: 10.1002/lary.21387. Epub 2011 Feb 4. PMID 21298638
- [Background] Pekala K, Chandra RK, Turner JH. Efficacy of olfactory training in patients with olfactory loss: a systematic review and meta-analysis. Int Forum Allergy Rhinol. 2016 Mar;6(3):299-307. doi: 10.1002/alr.21669. Epub 2015 Dec 1. PMID 26624966
- [Background] Doty RL. Olfaction in Parkinson's disease and related disorders. Neurobiol Dis. 2012 Jun;46(3):527-52. doi: 10.1016/j.nbd.2011.10.026. Epub 2011 Dec 20. PMID 22192366
- [Background] Boesveldt S, Postma EM, Boak D, Welge-Luessen A, Schopf V, Mainland JD, Martens J, Ngai J, Duffy VB. Anosmia-A Clinical Review. Chem Senses. 2017 Sep 1;42(7):513-523. doi: 10.1093/chemse/bjx025. PMID 28531300
- [Background] Hummel T, Rissom K, Reden J, Hahner A, Weidenbecher M, Huttenbrink KB. Effects of olfactory training in patients with olfactory loss. Laryngoscope. 2009 Mar;119(3):496-9. doi: 10.1002/lary.20101. PMID 19235739
- [Background] Konstantinidis I, Tsakiropoulou E, Bekiaridou P, Kazantzidou C, Constantinidis J. Use of olfactory training in post-traumatic and postinfectious olfactory dysfunction. Laryngoscope. 2013 Dec;123(12):E85-90. doi: 10.1002/lary.24390. Epub 2013 Oct 4. PMID 24114690
- [Background] Kollndorfer K, Fischmeister FP, Kowalczyk K, Hoche E, Mueller CA, Trattnig S, Schopf V. Olfactory training induces changes in regional functional connectivity in patients with long-term smell loss. Neuroimage Clin. 2015 Sep 15;9:401-10. doi: 10.1016/j.nicl.2015.09.004. eCollection 2015. PMID 26594622
- [Background] Kollndorfer K, Kowalczyk K, Hoche E, Mueller CA, Pollak M, Trattnig S, Schopf V. Recovery of olfactory function induces neuroplasticity effects in patients with smell loss. Neural Plast. 2014;2014:140419. doi: 10.1155/2014/140419. Epub 2014 Dec 3. PMID 25544900
- [Background] Wang L, Chen L, Jacob T. Evidence for peripheral plasticity in human odour response. J Physiol. 2004 Jan 1;554(Pt 1):236-44. doi: 10.1113/jphysiol.2003.054726. PMID 14678505
- [Background] Gudziol V, Lotsch J, Hahner A, Zahnert T, Hummel T. Clinical significance of results from olfactory testing. Laryngoscope. 2006 Oct;116(10):1858-63. doi: 10.1097/01.mlg.0000234915.51189.cb. PMID 17003712
- [Background] Doty RL, Shaman P, Dann M. Development of the University of Pennsylvania Smell Identification Test: a standardized microencapsulated test of olfactory function. Physiol Behav. 1984 Mar;32(3):489-502. doi: 10.1016/0031-9384(84)90269-5. PMID 6463130
- [Background] Doty RL. Office procedures for quantitative assessment of olfactory function. Am J Rhinol. 2007 Jul-Aug;21(4):460-73. doi: 10.2500/ajr.2007.21.3043. PMID 17882917
- [Background] Doty RL, Frye RE, Agrawal U. Internal consistency reliability of the fractionated and whole University of Pennsylvania Smell Identification Test. Percept Psychophys. 1989 May;45(5):381-4. doi: 10.3758/bf03210709. PMID 2726398
- [Background] Hummel C, Zucco GM, Iannilli E, Maboshe W, Landis BN, Hummel T. OLAF: standardization of international olfactory tests. Eur Arch Otorhinolaryngol. 2012 Mar;269(3):871-80. doi: 10.1007/s00405-011-1770-0. Epub 2011 Sep 21. PMID 21935630
- [Background] Marine N, Boriana A. Olfactory markers of depression and Alzheimer's disease. Neurosci Biobehav Rev. 2014 Sep;45:262-70. doi: 10.1016/j.neubiorev.2014.06.016. Epub 2014 Jul 6. PMID 25003804
- [Background] Doty RL. Olfactory dysfunction and its measurement in the clinic. World J Otorhinolaryngol Head Neck Surg. 2015 Oct 26;1(1):28-33. doi: 10.1016/j.wjorl.2015.09.007. eCollection 2015 Sep. PMID 29204537
- [Background] Hugh SC, Siu J, Hummel T, Forte V, Campisi P, Papsin BC, Propst EJ. Olfactory testing in children using objective tools: comparison of Sniffin' Sticks and University of Pennsylvania Smell Identification Test (UPSIT). J Otolaryngol Head Neck Surg. 2015 Mar 1;44(1):10. doi: 10.1186/s40463-015-0061-y. PMID 25890082
- [Background] Dunlop BW, Gray J, Rapaport MH. Transdiagnostic Clinical Global Impression Scoring for Routine Clinical Settings. Behav Sci (Basel). 2017 Jun 27;7(3):40. doi: 10.3390/bs7030040. PMID 28653978
- [Background] Frasnelli J, Hummel T. Olfactory dysfunction and daily life. Eur Arch Otorhinolaryngol. 2005 Mar;262(3):231-5. doi: 10.1007/s00405-004-0796-y. Epub 2004 May 5. PMID 15133691
- [Background] Geissler K, Reimann H, Gudziol H, Bitter T, Guntinas-Lichius O. Olfactory training for patients with olfactory loss after upper respiratory tract infections. Eur Arch Otorhinolaryngol. 2014 Jun;271(6):1557-62. doi: 10.1007/s00405-013-2747-y. Epub 2013 Oct 6. PMID 24096819
- [Background] Albrecht J, Anzinger A, Kopietz R, Schopf V, Kleemann AM, Pollatos O, Wiesmann M. Test-retest reliability of the olfactory detection threshold test of the Sniffin' sticks. Chem Senses. 2008 Jun;33(5):461-7. doi: 10.1093/chemse/bjn013. Epub 2008 Apr 4. PMID 18390818
- [Background] Fleiner F, Lau L, Goktas O. Active olfactory training for the treatment of smelling disorders. Ear Nose Throat J. 2012 May;91(5):198-203, 215. doi: 10.1177/014556131209100508. PMID 22614554
- [Background] Kawase T, Sakamoto S, Hori Y, Maki A, Suzuki Y, Kobayashi T. Bimodal audio-visual training enhances auditory adaptation process. Neuroreport. 2009 Sep 23;20(14):1231-4. doi: 10.1097/WNR.0b013e32832fbef8. PMID 19629016
- [Background] Isaiah A, Vongpaisal T, King AJ, Hartley DE. Multisensory training improves auditory spatial processing following bilateral cochlear implantation. J Neurosci. 2014 Aug 13;34(33):11119-30. doi: 10.1523/JNEUROSCI.4767-13.2014. PMID 25122908
- [Background] Bavelier D, Dye MW, Hauser PC. Do deaf individuals see better? Trends Cogn Sci. 2006 Nov;10(11):512-8. doi: 10.1016/j.tics.2006.09.006. Epub 2006 Oct 2. PMID 17015029
- [Background] Hoffman HJ, Rawal S, Li CM, Duffy VB. New chemosensory component in the U.S. National Health and Nutrition Examination Survey (NHANES): first-year results for measured olfactory dysfunction. Rev Endocr Metab Disord. 2016 Jun;17(2):221-40. doi: 10.1007/s11154-016-9364-1. PMID 27287364
- [Background] Seiden AM, Duncan HJ. The diagnosis of a conductive olfactory loss. Laryngoscope. 2001 Jan;111(1):9-14. doi: 10.1097/00005537-200101000-00002. PMID 11192906
- [Background] Cain WS, Gent JF, Goodspeed RB, Leonard G. Evaluation of olfactory dysfunction in the Connecticut Chemosensory Clinical Research Center. Laryngoscope. 1988 Jan;98(1):83-8. doi: 10.1288/00005537-198801000-00017. PMID 3336267
- [Background] Deems DA, Doty RL, Settle RG, Moore-Gillon V, Shaman P, Mester AF, Kimmelman CP, Brightman VJ, Snow JB Jr. Smell and taste disorders, a study of 750 patients from the University of Pennsylvania Smell and Taste Center. Arch Otolaryngol Head Neck Surg. 1991 May;117(5):519-28. doi: 10.1001/archotol.1991.01870170065015. PMID 2021470
- [Background] Quint C, Temmel AF, Schickinger B, Pabinger S, Ramberger P, Hummel T. Patterns of non-conductive olfactory disorders in eastern Austria: a study of 120 patients from the Department of Otorhinolaryngology at the University of Vienna. Wien Klin Wochenschr. 2001 Jan 15;113(1-2):52-7. PMID 11233469
- [Background] Seiden AM. Postviral olfactory loss. Otolaryngol Clin North Am. 2004 Dec;37(6):1159-66. doi: 10.1016/j.otc.2004.06.007. PMID 15563908
- [Background] Suzuki M, Saito K, Min WP, Vladau C, Toida K, Itoh H, Murakami S. Identification of viruses in patients with postviral olfactory dysfunction. Laryngoscope. 2007 Feb;117(2):272-7. doi: 10.1097/01.mlg.0000249922.37381.1e. PMID 17277621
- [Background] Hedner M, Larsson M, Arnold N, Zucco GM, Hummel T. Cognitive factors in odor detection, odor discrimination, and odor identification tasks. J Clin Exp Neuropsychol. 2010 Dec;32(10):1062-7. doi: 10.1080/13803391003683070. Epub 2010 Apr 30. PMID 20437286
- [Background] Giacomelli A, Pezzati L, Conti F, Bernacchia D, Siano M, Oreni L, Rusconi S, Gervasoni C, Ridolfo AL, Rizzardini G, Antinori S, Galli M. Self-reported Olfactory and Taste Disorders in Patients With Severe Acute Respiratory Coronavirus 2 Infection: A Cross-sectional Study. Clin Infect Dis. 2020 Jul 28;71(15):889-890. doi: 10.1093/cid/ciaa330. No abstract available. PMID 32215618
- [Background] Lechien JR, Chiesa-Estomba CM, De Siati DR, Horoi M, Le Bon SD, Rodriguez A, Dequanter D, Blecic S, El Afia F, Distinguin L, Chekkoury-Idrissi Y, Hans S, Delgado IL, Calvo-Henriquez C, Lavigne P, Falanga C, Barillari MR, Cammaroto G, Khalife M, Leich P, Souchay C, Rossi C, Journe F, Hsieh J, Edjlali M, Carlier R, Ris L, Lovato A, De Filippis C, Coppee F, Fakhry N, Ayad T, Saussez S. Olfactory and gustatory dysfunctions as a clinical presentation of mild-to-moderate forms of the coronavirus disease (COVID-19): a multicenter European study. Eur Arch Otorhinolaryngol. 2020 Aug;277(8):2251-2261. doi: 10.1007/s00405-020-05965-1. Epub 2020 Apr 6. PMID 32253535
- [Background] Harless L, Liang J. Pharmacologic treatment for postviral olfactory dysfunction: a systematic review. Int Forum Allergy Rhinol. 2016 Jul;6(7):760-7. doi: 10.1002/alr.21727. Epub 2016 Feb 16. PMID 26879592
- [Derived] Khan AM, Piccirillo J, Kallogjeri D, Piccirillo JF. Efficacy of Combined Visual-Olfactory Training With Patient-Preferred Scents as Treatment for Patients With COVID-19 Resultant Olfactory Loss: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2023 Feb 1;149(2):141-149. doi: 10.1001/jamaoto.2022.4112. PMID 36580304
- See also: Official study web application for administration of smell training intervention. All study participants will receive login credentials. — https://outcomesresearch.github.io/volt